CLINICAL TRIAL: NCT07024394
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of Ruvometinib Tablets (FCN-159 Tablets) in Pediatric Participants With Neurofibromatosis Type 1
Brief Title: Follow-up Study to Evaluate the Safety and Efficacy of FCN-159 in Pediatric Participants With Neurofibromatosis Type 1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-002-LT
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FCN-159 (Experimental): Study Drug: FCN-159 Dosing Regimen: FCN-159 to be administered once daily until disease progression or study completion, whichever occurs first
  Interventions: Drug: Luvometinib Tablets

INTERVENTIONS:
Drug: Luvometinib Tablets — 5mg/m² (Maximum dose does not exceed 8mg, the recommended oral dose for adults), orally, once daily, until disease progression or study completion, whichever occurs first
  Other Names: FCN-159

SUMMARY:
FCN-159 (Luvometinib Tablets), an orally available and highly potent selective inhibitor of MEK1/2,demonstrated good tolerability and exhibited notable anti-tumor activity in pediatric pts with NF1-related PN in study NCT04954001.This study is a 5-year long-term follow-up of the FCN-159-002 study, involving all enrolled patients to further assess safety, growth and development effects, and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients from the pediatric cohort of the FCN-159-002 study. Willing to participate in the long-term follow-up study and capable of understanding and voluntarily signing the informed consent form.

Exclusion Criteria:

Any clinically significant condition that, in the investigator's judgment, may interfere with study participation or compliance with safety requirements.

Patients unable to comply with visit-related requirements.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-06-12 (Estimated); Primary Completion 2029-09-23 (Estimated); Study Completion 2029-09-23 (Estimated)

PRIMARY OUTCOMES:
long term safty | Through study completion, about 5 years
  Adverse events during treatment of FCN-159 will be assessed by the investigators according to CTCAE 5.0.

SECONDARY OUTCOMES:
Height in centimeters | Through study completion, about 5 years
  Height will be measured in centimeters, with subsequent plotting of height growth curves and calculation of growth velocity.
Weight in kilograms | Through study completion, about 5 years
  Weight will be measured in kilograms, with subsequent plotting of weight growth curves.
Tanner stage | Through study completion, about 5 years
  Tanner stage will be examined, and the mean age for each Tanner stage will be calculated.
Progression-Free Survival (PFS) | Through study completion, about 5 years
  PFS assessed per REiNS (Response Evaluation in Neurofibromatosis and Schwannomatosis) criteria by inverstigator
Objective response rate (ORR) | Through study completion, about 5 years
  ORR assessed per REiNS (Response Evaluation in Neurofibromatosis and Schwannomatosis) criteria by inverstigator.
Changes in pain intensity | Through study completion, about 5 years
  Changes in pain intensity score relative to baseline will be assessed according to 11-point Numerical Rating Scale (NRS-11).NRS-11 quantifies pain intensity on a scale from 0 to 10, 0 represents "No pain" ,10 represents "The worst pain imaginable".

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China